CLINICAL TRIAL: NCT02129387
Title: EEG & Behavioral Predictors of Changes in Smoking Trajectories in Young Light Smokers
Status: Completed | Type: Observational
Sponsor: Southern Illinois University Carbondale (Other)
Responsible Party: Sponsor
Other Study IDs: 1R01DA036032-01 (NIH)
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Nicotine Dependence
Keywords: Nicotine; Smoking Progression; EEG; Young adults; Light smokers; rs1051730 genotype
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, saliva
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the proposal is to identify new predictors of smoking progression in young light smokers (YLS: 18-25 years & cpd < 5) using an 18-month longitudinal design and to relate these predictors of progression to the genetic profile most highly associated with smoking progression. A number of novel predictors will be assessed in 128 YLS. Predictors will include individual differences (IDs) in EEG, reward sensitivity, attentional performance, and mood during abstinence and in response to standardized and to self-selected acute nicotine doses (ANIC), as well as genetically influenced affective traits, and smoking history. The associations of a compelling genetic functional variant polymorphism, rs16969968, in the alpha5 nicotinic receptor subunit will also be related to smoking progression and the novel predictors. The study is expected to provide insights into IDs in mechanisms and predictors that contribute to smoking trajectories in YLS and thereby lead to targeted pharmacotherapy and behavioral interventions for at-risk YLS.

DETAILED DESCRIPTION:
The purpose of the proposal is to identify new biobehavioral endophenotypes that predict smoking progression in young light smokers (YLS: 18-25 years & cpd < 5) using an 18-month longitudinal design and to relate these endophenotypes and progression to the genetic profile most highly associated with smoking progression. A number of novel predictors will be assessed in 128 YLS. Predictors will include individual differences (IDs) in EEG, reward sensitivity, attentional performance, and mood during abstinence and in response to standardized and to self-selected acute nicotine doses (ANIC), as well as genetically influenced affective traits, and smoking history. The associations of a compelling genetic functional variant polymorphism, rs16969968, in the alpha5 nicotinic receptor subunit will also be related to smoking progression and the novel predictors. The study is expected to provide insights into IDs in mechanisms and endophenotypes that contribute to smoking trajectories in YLS and thereby lead to targeted pharmacotherapy and behavioral interventions for at-risk YLS.

ELIGIBILITY:
Inclusion Criteria:

* smokers of 3 to 30 cigarettes per week for past 6 months

Exclusion Criteria:

* Smoking fewer than 3 or more than 30 tobacco cigarettes per week
* Never smoked more than 30 cigarettes per week
* Psychoactive drug use other than caffeine or occasional marijuana
* Current serious psychiatric diagnosis (e.g., major depressive disorder)
* Recent drug dependence
* Left-handed
* Color blind

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample of young light smokers
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
change in smoking and salivary cotinine concentration | 18 months
  Change in smoking and salivary cotinine concentration from baseline to 18 months will be assessed at 3 month intervals-- 3, 6, 9, 12, 15, and 18 months after initial assessments.

SECONDARY OUTCOMES:
reason for change in smoke rate | 18 months after initial assessment
  Self-reported reasons for changing smoking or for continuing to smoke at the same rate will be assessed a 3-month intervals until 18 months after baseline assessment.

CONTACTS AND LOCATIONS:
Overall Officials: David G Gilbert, PhD, Principal Investigator — Southern Illinois University Carbondale
Locations (1):
- Southern Illinois University Carbondale Department of Psychology, Carbondale, Illinois, United States

REFERENCES:
- [Derived] Gunn MP, Rose GM, Whitton AE, Pizzagalli DA, Gilbert DG. Smoking Progression and Nicotine-Enhanced Reward Sensitivity Predicted by Resting-State Functional Connectivity in Salience and Executive Control Networks. Nicotine Tob Res. 2024 Sep 23;26(10):1305-1312. doi: 10.1093/ntr/ntae084. PMID 38624067
- [Derived] Whitton AE, Rabinovich NE, Lindt JD, Pergadia ML, Pizzagalli DA, Gilbert DG. Genetic and Depressive Traits Moderate the Reward-Enhancing Effects of Acute Nicotine in Young Light Smokers. Nicotine Tob Res. 2021 Aug 29;23(10):1779-1786. doi: 10.1093/ntr/ntab072. PMID 33844007